CLINICAL TRIAL: NCT00235443
Title: A Multi-Center, Open-Label, Follow-On Trial to Assess the Long Term Safety and Efficacy of SPM 927 in Subjects With Painful Distal Diabetic Neuropathy
Brief Title: A Follow-On Trial to Assess the Long Term Safety and Efficacy of SPM 927 in Painful Distal Diabetic Neuropathy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0745
Expanded Access: NCT03559673 (No longer available)
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Results first posted 2009-10-05 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2017-07

CONDITIONS: Diabetic Neuropathy
Keywords: Painful Distal Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Lacosamide; 2-(acetylamino)-3-methoxy-N-(phenylmethyl)-, (2R)-

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Open label doses (two times per day) include 100mg/day, 200mg/day, 300mg/day, 400mg/day, 500mg/day, 600mg/day
  Interventions: Drug: lacosamide

INTERVENTIONS:
Drug: lacosamide — Open-label treatment (two times per day) with film-coated tablets include 100mg/day, 200mg/day, 300mg/day, 400mg/day, 500mg/day, and 600mg/day throughout individual study period.
  Other Names: SPM927

SUMMARY:
Phase 2/3 open-label trial to assess the safety and tolerability of long-term treatment with lacosamide (SPM 927) in subjects with painful diabetic neuropathy. The safety and tolerability of the different doses of lacosamide will be investigated.

DETAILED DESCRIPTION:
This phase 2/3 open-label trial is being conducted at approximately 100 sites in the US to assess the safety and tolerability of long-term treatment with lacosamide (SPM 927) in subjects with painful diabetic neuropathy. Approximately 525 subjects will be enrolled. To qualify for this trial, subjects with symptoms of painful distal diabetic neuropathy ranging in duration from 6 months to 5 years must have completed trials SP665, SP742, or SP768 and, in the investigator's opinion, may benefit from long-term administration of lacosamide. Subjects will be titrated to their optimal dose of lacosamide (up to 600mg/day). The safety and tolerability of the different doses of lacosamide will be investigated throughout the trial. In addition, to determine what effect lacosamide has on diabetic neuropathic pain, subjects will use a diary to record their daily pain intensity and pain interference with sleep and activity. Subjects' quality of life will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who completed Study SP665, SP742, or SP768 and, in the investigators opinion, might benefit from long-term administration of SPM 927. Exception: subjects who prematurely discontinued Study SP742 or SP768 due to lack of efficacy or due to intolerability to trial medication may be eligible to participate in Study SP745, after consultation with the medical monitor.

Exclusion Criteria:

* Subject has clinically relevant electrocardiogram (ECG) abnormalities, or QT-corrected (QTc) interval >=500 milliseconds (ms), and/or a QTc interval increase of >=60ms from the mean pre-dose QTc value at Visit 2 of Studies SP665, SP742 or SP768.
* Subject has aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >=3 times the upper limit of the normal range (ULN) with total bilirubin >=2 times ULN or transaminases (AST and/or ALT) >=5 times ULN.
* Subject has a clinically relevant medical condition that, in the opinion of the investigator, jeopardizes or compromises the subject's ability to participate in this trial.

Ages: 32 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2004-09; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (84):
- United States (84):
  - Anniston, Alabama
  - Hoover, Alabama
  - Huntsville, Alabama
  - Northport, Alabama
  - Tuscaloosa, Alabama
  - Peoria, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Hot Springs, Arkansas
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Irvine, California
  - Los Angeles, California
  - San Diego, California
  - Santa Monica, California
  - Spring Valley, California
  - Tustin, California
  - Walnut Creek, California
  - Denver, Colorado
  - Stratford, Connecticut
  - Newark, Delaware
  - Wilmington, Delaware
  - Bradenton, Florida
  - Clearwater, Florida
  - Fort Myers, Florida
  - New Port Richey, Florida
  - Ocala, Florida
  - Pembroke Pines, Florida
  - Pinellas Park, Florida
  - South Miami, Florida
  - St. Petersburg, Florida
  - Sunrise, Florida
  - Tallahassee, Florida
  - Marietta, Georgia
  - Chicago, Illinois
  - Elk Grove Village, Illinois
  - North Chicago, Illinois
  - Evansville, Indiana
  - West Des Moines, Iowa
  - Crestview Hills, Kentucky
  - Louisville, Kentucky
  - Madisonville, Kentucky
  - Paducah, Kentucky
  - Owings Mills, Maryland
  - Towson, Maryland
  - Brockton, Massachusetts
  - Ann Arbor, Michigan
  - St Louis, Missouri
  - Great Falls, Montana
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Lawrenceville, New Jersey
  - Voorhees Township, New Jersey
  - Albany, New York
  - Mineola, New York
  - White Plains, New York
  - Charlotte, North Carolina
  - Greensboro, North Carolina
  - Greenville, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Medford, Oregon
  - Portland, Oregon
  - Upland, Pennsylvania
  - Greer, South Carolina
  - Bristol, Tennessee
  - Nashville, Tennessee
  - Amarillo, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Richardson, Texas
  - San Antonio, Texas
  - Bennington, Vermont
  - Richmond, Virginia
  - Salem, Virginia
  - Virginia Beach, Virginia
  - Spokane, Washington
  - Tacoma, Washington
  - Wenatchee, Washington

REFERENCES:
- [Derived] Shaibani A, Biton V, Rauck R, Koch B, Simpson J. Long-term oral lacosamide in painful diabetic neuropathy: a two-year open-label extension trial. Eur J Pain. 2009 May;13(5):458-63. doi: 10.1016/j.ejpain.2008.05.016. Epub 2008 Jul 10. PMID 18619874
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial SP745 (NCT00235443) was conducted in 93 sites in the US and 89 of these sites screened at least 1 subject. The first subject was enrolled on 13Sep2004 and the last subject completed on 25Jul2008.
Groups:
- Lacosamide 100mg/Day; Lacosamide 200mg/Day; Lacosamide 300mg/Day; Lacosamide 400mg/Day; Lacosamide 500mg/Day; Lacosamide 600mg/Day: Modal dose = Open label doses (two times per day) include 100mg/day, 200mg/day, 300mg/day, 400mg/day, 500mg/day, 600mg/day
Period: Overall Study
Arm/Group | Lacosamide 100mg/Day | Lacosamide 200mg/Day | Lacosamide 300mg/Day | Lacosamide 400mg/Day | Lacosamide 500mg/Day | Lacosamide 600mg/Day
Started | 11 | 57 | 85 | 205 | 39 | 54
Completed | 3 | 19 | 23 | 108 | 9 | 9
Not Completed | 8 | 38 | 62 | 97 | 30 | 45
Not completed — Adverse Event | 4 | 12 | 17 | 44 | 10 | 15
Not completed — Lack of Efficacy | 0 | 1 | 5 | 12 | 2 | 9
Not completed — Withdrawal by Subject | 3 | 9 | 25 | 24 | 10 | 12
Not completed — Lost to Follow-up | 0 | 8 | 6 | 6 | 4 | 3
Not completed — Unsatisfactory compliance | 0 | 2 | 3 | 4 | 1 | 0
Not completed — Other reasons for premature termination | 1 | 6 | 6 | 7 | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lacosamide 100mg/Day | Lacosamide 200mg/Day | Lacosamide 300mg/Day | Lacosamide 400mg/Day | Lacosamide 500mg/Day | Lacosamide 600mg/Day | Total
Number analyzed (Participants) | 11 | 57 | 85 | 205 | 39 | 54 | 451
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 38 | 61 | 160 | 30 | 44 | 339
  >=65 years | 5 | 19 | 24 | 45 | 9 | 10 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (8.16) | 59.3 (10.53) | 60.5 (8.55) | 57.3 (9.43) | 56.9 (9.52) | 55.5 (10.10) | 58.1 (9.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 33 | 48 | 80 | 16 | 18 | 200
  Male | 6 | 24 | 37 | 125 | 23 | 36 | 251
Region of Enrollment [Number; unit: participants]
  United States | 11 | 57 | 85 | 205 | 39 | 54 | 451

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events (AEs) Reported Spontaneously by the Subject or Observed by the Investigator.
Description: Number of subjects with adverse events (AEs) reported spontaneously by the subject or observed by the investigator (serious and non-serious).
Time Frame: Throughout the study up to a maximum study period of 2.8 years
Population: Safety population are subjects who took at least one dose of lacosamide (LCM).
Measure: Number; unit: Participants
Groups:
- Total: All modal dose groups combined
Arm/Group | Lacosamide 100mg/Day | Lacosamide 200mg/Day | Lacosamide 300mg/Day | Lacosamide 400mg/Day | Lacosamide 500mg/Day | Lacosamide 600mg/Day | Total
Number analyzed (Participants) | 11 | 57 | 85 | 205 | 39 | 54 | 451
Participants | 11 | 52 | 74 | 196 | 33 | 50 | 416

2. Secondary Outcome: Change From Baseline in Average Daily Pain Score Using an 11-point Likert Scale (0-10).
Description: Change from Baseline in average daily pain score using an 11-point Likert scale (0-10). On Likert scale, 0=no pain and 10=worst possible pain.
Time Frame: Baseline to end of entire treatment phase (maximum study period of 2.8 years).
Population: Safety population are subjects who took at least one dose of lacosamide (LCM).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lacosamide 100mg/Day | Lacosamide 200mg/Day | Lacosamide 300mg/Day | Lacosamide 400mg/Day | Lacosamide 500mg/Day | Lacosamide 600mg/Day | Total
Number analyzed (Participants) | 11 | 56 | 80 | 204 | 38 | 53 | 442
Units on a scale | -5.15 (2.345) | -4.30 (1.991) | -3.70 (2.020) | -3.29 (1.872) | -3.54 (1.602) | -2.73 (2.064) | -3.49 (1.982)

3. Secondary Outcome: Change From Baseline in Average Pain Score as Measured by a 100mm Visual Analogue Scale (VAS).
Description: Change from Baseline in average pain score as measured by a 100mm Visual Analogue Scale (VAS). On VAS 0mm=no pain and 100mm=worst possible pain.
Time Frame: Baseline to end of entire treatment phase (maximum study period of 2.8 years).
Population: Safety population are subjects who took at least one dose of lacosamide (LCM).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lacosamide 100mg/Day | Lacosamide 200mg/Day | Lacosamide 300mg/Day | Lacosamide 400mg/Day | Lacosamide 500mg/Day | Lacosamide 600mg/Day | Total
Number analyzed (Participants) | 11 | 57 | 81 | 205 | 39 | 54 | 447
Units on a scale | -47.83 (34.022) | -43.06 (23.901) | -35.24 (26.837) | -30.06 (23.723) | -36.73 (18.025) | -27.70 (22.427) | -33.39 (24.484)

4. Secondary Outcome: Patient's Global Impression of Change (PGIC) From Baseline in Pain.
Description: Patient's Global Impression of Change (PGIC) from Baseline in Pain. Original categorical responses are much worse, moderately worse, mildly worst, no change, mildly better, moderately better, and much better. Reported results are presented as Better (sum of mildly, moderately, or much better), No Change, or Worse (sum of mildly, moderately, or much worse).
Time Frame: Baseline to Termination Visit
Population: Safety population are subjects who took at least one dose of lacosamide (LCM).
Measure: Number; unit: Participants
Arm/Group | Lacosamide 100mg/Day | Lacosamide 200mg/Day | Lacosamide 300mg/Day | Lacosamide 400mg/Day | Lacosamide 500mg/Day | Lacosamide 600mg/Day | Total
Number analyzed (Participants) | 11 | 45 | 62 | 182 | 30 | 42 | 372
Participants
  Better | 10 | 42 | 50 | 147 | 26 | 34 | 309
  No Change | 0 | 3 | 10 | 15 | 0 | 1 | 29
  Worse | 1 | 0 | 2 | 20 | 4 | 7 | 34

5. Secondary Outcome: Within-subject Change in Neuropathic Pain Using the Neuropathic Pain Scale (NPS) - Intensity.
Description: Within-subject change in neuropathic pain using the Neuropathic Pain Scale (NPS) for intensity of pain where 0=no pain and 10=most intense pain sensation imaginable.
Time Frame: Baseline to Termination Visit
Population: Safety population are subjects who took at least one dose of lacosamide (LCM).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lacosamide 100mg/Day | Lacosamide 200mg/Day | Lacosamide 300mg/Day | Lacosamide 400mg/Day | Lacosamide 500mg/Day | Lacosamide 600mg/Day | Total
Number analyzed (Participants) | 10 | 45 | 62 | 181 | 30 | 42 | 370
Units on a scale | -4.6 (2.63) | -4.4 (3.03) | -3.1 (2.86) | -2.7 (2.96) | -3.5 (2.22) | -2.0 (2.61) | -3.0 (2.92)

6. Secondary Outcome: Within-subject Change in Neuropathic Pain Using the Neuropathic Pain Scale (NPS) - Sharpness
Description: Within-subject change in neuropathic pain using the Neuropathic Pain Scale (NPS) for sharpness of pain where 0=not sharp and 10=most sharp sensation imaginable ("like a knife").
Time Frame: Baseline to Termination Visit
Population: Safety population are subjects who took at least one dose of lacosamide (LCM).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lacosamide 100mg/Day | Lacosamide 200mg/Day | Lacosamide 300mg/Day | Lacosamide 400mg/Day | Lacosamide 500mg/Day | Lacosamide 600mg/Day | Total
Number analyzed (Participants) | 10 | 45 | 62 | 181 | 30 | 42 | 370
Units on a scale | -4.5 (2.76) | -4.2 (3.07) | -3.3 (3.25) | -2.8 (3.20) | -3.9 (2.51) | -1.9 (3.00) | -3.1 (3.17)

7. Secondary Outcome: Within-subject Change in Neuropathic Pain Using the Neuropathic Pain Scale (NPS) - Heat
Description: Within-subject change in neuropathic pain using the Neuropathic Pain Scale (NPS) with heat sensation where 0=not hot and 10=the most hot sensation imaginable ("on fire").
Time Frame: Baseline to Termination Visit
Population: Safety population are subjects who took at least one dose of lacosamide (LCM).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lacosamide 100mg/Day | Lacosamide 200mg/Day | Lacosamide 300mg/Day | Lacosamide 400mg/Day | Lacosamide 500mg/Day | Lacosamide 600mg/Day | Total
Number analyzed (Participants) | 10 | 45 | 62 | 181 | 30 | 42 | 370
Units on a scale | -5.3 (3.74) | -3.0 (3.65) | -3.1 (3.44) | -2.6 (3.14) | -2.8 (2.58) | -1.2 (2.86) | -2.7 (3.26)

8. Secondary Outcome: Within-subject Change in Neuropathic Pain Using the Neuropathic Pain Scale (NPS) - Dullness
Description: Within-subject change in neuropathic pain using the Neuropathic Pain Scale (NPS) with dullness of pain where 0=not dull and 10=most dull sensation imaginable.
Time Frame: Baseline to Termination Visit
Population: Safety population are subjects who took at least one dose of lacosamide (LCM).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lacosamide 100mg/Day | Lacosamide 200mg/Day | Lacosamide 300mg/Day | Lacosamide 400mg/Day | Lacosamide 500mg/Day | Lacosamide 600mg/Day | Total
Number analyzed (Participants) | 10 | 45 | 62 | 181 | 30 | 42 | 370
Units on a scale | -3.4 (2.41) | -2.6 (3.03) | -2.6 (2.88) | -2.4 (3.34) | -2.4 (3.65) | -1.8 (3.23) | -2.4 (3.22)

9. Secondary Outcome: Within-subject Change in Neuropathic Pain Using the Neuropathic Pain Scale (NPS) - Cold
Description: Within-subject change in neuropathic pain using the Neuropathic Pain Scale (NPS) with cold sensation where 0=not cold and 10=most cold sensation imaginable ("freezing").
Time Frame: Baseline to Termination Visit
Population: Safety population are subjects who took at least one dose of lacosamide (LCM).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lacosamide 100mg/Day | Lacosamide 200mg/Day | Lacosamide 300mg/Day | Lacosamide 400mg/Day | Lacosamide 500mg/Day | Lacosamide 600mg/Day | Total
Number analyzed (Participants) | 10 | 45 | 61 | 180 | 30 | 42 | 368
Units on a scale | -1.6 (3.34) | -1.9 (3.14) | -1.2 (3.13) | -1.7 (3.19) | -2.2 (3.64) | -0.5 (3.01) | -1.5 (3.20)

10. Secondary Outcome: Within-subject Change in Neuropathic Pain Using the Neuropathic Pain Scale (NPS) - Sensitivity
Description: Within-subject change in neuropathic pain using the Neuropathic Pain Scale (NPS) with sensitivity of pain where 0=not sensitive and 10=most sensitive sensation imaginable ("raw skin").
Time Frame: Baseline to Termination Visit
Population: Safety population are subjects who took at least one dose of lacosamide (LCM).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lacosamide 100mg/Day | Lacosamide 200mg/Day | Lacosamide 300mg/Day | Lacosamide 400mg/Day | Lacosamide 500mg/Day | Lacosamide 600mg/Day | Total
Number analyzed (Participants) | 10 | 45 | 61 | 181 | 30 | 42 | 369
Units on a scale | -2.8 (4.78) | -3.4 (3.46) | -1.8 (3.10) | -2.1 (3.44) | -2.7 (3.24) | -1.4 (3.26) | -2.2 (3.42)

11. Secondary Outcome: Within-subject Change in Neuropathic Pain Using the Neuropathic Pain Scale (NPS) - Itchiness
Description: Within-subject change in neuropathic pain using the Neuropathic Pain Scale (NPS) with itchiness where 0=not itchy and 10=most itchy sensation imaginable ("like poison oak").
Time Frame: Baseline to Termination Visit
Population: Safety population are subjects who took at least one dose of lacosamide (LCM).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lacosamide 100mg/Day | Lacosamide 200mg/Day | Lacosamide 300mg/Day | Lacosamide 400mg/Day | Lacosamide 500mg/Day | Lacosamide 600mg/Day | Total
Number analyzed (Participants) | 10 | 45 | 61 | 181 | 30 | 42 | 369
Units on a scale | -2.2 (2.94) | -2.0 (3.19) | -1.4 (3.26) | -1.1 (3.03) | -2.1 (2.57) | -0.5 (2.79) | -1.3 (3.05)

12. Secondary Outcome: Within-subject Change in Neuropathic Pain Using the Neuropathic Pain Scale (NPS) - Unpleasantness
Description: Within-subject change in neuropathic pain using the Neuropathic Pain Scale (NPS) with unpleasantness where 0=not pleasant and 10=most unpleasant sensation imaginable ("intolerable").
Time Frame: Baseline to Termination Visit
Population: Safety population are subjects who took at least one dose of lacosamide (LCM).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lacosamide 100mg/Day | Lacosamide 200mg/Day | Lacosamide 300mg/Day | Lacosamide 400mg/Day | Lacosamide 500mg/Day | Lacosamide 600mg/Day | Total
Number analyzed (Participants) | 10 | 45 | 61 | 180 | 30 | 42 | 368
Units on a scale | -5.0 (3.56) | -4.0 (3.15) | -3.3 (3.08) | -2.9 (2.96) | -3.3 (2.85) | -1.5 (2.61) | -3.0 (3.04)

13. Secondary Outcome: Within-subject Change in Neuropathic Pain Using the Neuropathic Pain Scale (NPS) - Deep Pain
Description: Within-subject change in neuropathic pain using the Neuropathic Pain Scale (NPS) with deep pain where 0=no deep pain and 10=most intense deep pain sensation imaginable.
Time Frame: Baseline to Termination Visit
Population: Safety population are subjects who took at least one dose of lacosamide (LCM).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lacosamide 100mg/Day | Lacosamide 200mg/Day | Lacosamide 300mg/Day | Lacosamide 400mg/Day | Lacosamide 500mg/Day | Lacosamide 600mg/Day | Total
Number analyzed (Participants) | 10 | 45 | 61 | 180 | 30 | 42 | 368
Units on a scale | -4.5 (3.34) | -3.3 (3.58) | -3.2 (3.35) | -2.7 (3.11) | -3.3 (2.94) | -1.5 (2.88) | -2.8 (3.21)

14. Secondary Outcome: Within-subject Change in Neuropathic Pain Using the Neuropathic Pain Scale (NPS) - Surface Pain
Description: Within-subject change in neuropathic pain using the Neuropathic Pain Scale (NPS) with surface pain where 0=no surface pain and 10=most intense surface pain imaginable.
Time Frame: Baseline to Termination Visit
Population: Safety population are subjects who took at least one dose of lacosamide (LCM).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lacosamide 100mg/Day | Lacosamide 200mg/Day | Lacosamide 300mg/Day | Lacosamide 400mg/Day | Lacosamide 500mg/Day | Lacosamide 600mg/Day | Total
Number analyzed (Participants) | 10 | 45 | 60 | 179 | 30 | 42 | 366
Units on a scale | -3.5 (4.30) | -3.3 (3.53) | -3.3 (3.28) | -2.6 (2.96) | -2.7 (2.89) | -1.5 (2.95) | -2.7 (3.15)

15. Secondary Outcome: Change From Baseline in Average Pain Interference With Sleep (11-point Likert Scale)
Description: Change from Baseline in average pain interference with sleep (11-point Likert scale) where 0=no interference with sleep and 10=worst possible interference with sleep.
Time Frame: Baseline to end of entire treatment phase visit
Population: Safety population are subjects who took at least one dose of lacosamide (LCM).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lacosamide 100mg/Day | Lacosamide 200mg/Day | Lacosamide 300mg/Day | Lacosamide 400mg/Day | Lacosamide 500mg/Day | Lacosamide 600mg/Day | Total
Number analyzed (Participants) | 11 | 56 | 80 | 203 | 38 | 53 | 441
Units on a scale | -4.62 (2.950) | -3.86 (2.050) | -3.32 (2.077) | -3.15 (2.150) | -3.34 (1.852) | -2.85 (2.427) | -3.29 (2.173)

16. Secondary Outcome: Change From Baseline in Average Pain Interference With Activity (11-point Likert Scale)
Description: Change from Baseline in average pain interference with activity (11-point Likert scale) where 0=no interfence with activity and 10=worst possible interference with activity.
Time Frame: Baseline to end of entire treatment phase visit
Population: Safety population are subjects who took at least one dose of lacosamide (LCM).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lacosamide 100mg/Day | Lacosamide 200mg/Day | Lacosamide 300mg/Day | Lacosamide 400mg/Day | Lacosamide 500mg/Day | Lacosamide 600mg/Day | Total
Number analyzed (Participants) | 11 | 56 | 80 | 203 | 38 | 53 | 441
Units on a scale | -4.82 (2.927) | -3.82 (2.185) | -3.36 (2.163) | -3.00 (2.038) | -3.30 (1.808) | -2.54 (2.261) | -3.18 (2.147)

17. Secondary Outcome: Change From Baseline in Quality of Life Using the SF-36 Health Survey - Physical Component Summary (PCS)
Description: Change from Baseline in quality of life using the SF-36 Health Survey - Physical Component Summary (PCS). Values range from 0 to 100 with high values indicating a good condition. Positive change in baseline values indicate improvement in quality of life.
Time Frame: Baseline to Termination Visit
Population: Safety population are subjects who took at least one dose of lacosamide (LCM).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lacosamide 100mg/Day | Lacosamide 200mg/Day | Lacosamide 300mg/Day | Lacosamide 400mg/Day | Lacosamide 500mg/Day | Lacosamide 600mg/Day | Total
Number analyzed (Participants) | 11 | 45 | 61 | 179 | 30 | 42 | 368
Units on a scale | 3.3 (11.25) | 5.5 (10.50) | 5.1 (9.14) | 3.7 (8.80) | 3.5 (6.70) | 2.1 (8.56) | 4.0 (8.98)

18. Secondary Outcome: Change From Baseline in Quality of Life Using the SF-36 Health Survey - Mental Component Summary (MCS)
Description: Change from Baseline in quality of life using the SF-36 Health Survey - Mental Component Summary (MCS). Values range from 0 to 100 with high values indicating a good condition. Positive change in baseline values indicate improvement in quality of life.
Time Frame: Baseline to Termination Visit
Population: Safety population are subjects who took at least one dose of lacosamide (LCM).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lacosamide 100mg/Day | Lacosamide 200mg/Day | Lacosamide 300mg/Day | Lacosamide 400mg/Day | Lacosamide 500mg/Day | Lacosamide 600mg/Day | Total
Number analyzed (Participants) | 11 | 45 | 61 | 179 | 30 | 42 | 368
Units on a scale | -3.4 (10.66) | -0.1 (12.60) | 0.7 (10.78) | -1.1 (11.09) | -3.7 (14.34) | -0.4 (12.02) | -0.9 (11.60)

ADVERSE EVENTS:
Time Frame: 3 years, 10 months
Arm/Group | Lacosamide 100mg/Day | Lacosamide 200mg/Day | Lacosamide 300mg/Day | Lacosamide 400mg/Day | Lacosamide 500mg/Day | Lacosamide 600mg/Day | Total
Serious Adverse Events (participants affected / at risk) | 1/11 | 13/57 | 17/85 | 52/205 | 10/39 | 7/54 | 100/451
Other Adverse Events (participants affected / at risk) | 10/11 | 47/57 | 68/85 | 183/205 | 28/39 | 43/54 | 379/451
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide 100mg/Day (N=11) | Lacosamide 200mg/Day (N=57) | Lacosamide 300mg/Day (N=85) | Lacosamide 400mg/Day (N=205) | Lacosamide 500mg/Day (N=39) | Lacosamide 600mg/Day (N=54) | Total (N=451)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 7 (7)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 3 (3)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Artioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal angiodysplasia haemorrhagic (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (2) | 5 (5) | 1 (1) | 1 (1) | 8 (9)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 4 (4)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis C antibody positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram PR prolongation (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diabetic foot (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 4 (4)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hodgkin's disease mixed cellularity stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inflammatory carcinoma of the breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Depression suicidal (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Toe amputation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Shoulder operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aortic dilatation (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide 100mg/Day (N=11) | Lacosamide 200mg/Day (N=57) | Lacosamide 300mg/Day (N=85) | Lacosamide 400mg/Day (N=205) | Lacosamide 500mg/Day (N=39) | Lacosamide 600mg/Day (N=54) | Total (N=451)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 4 (4) | 10 (10) | 1 (1) | 1 (1) | 18 (18)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 4 (5)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 3 (3) | 2 (5) | 8 (9) | 1 (1) | 3 (3) | 17 (21)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 3 (3) | 11 (12) | 1 (1) | 2 (2) | 17 (18)
Cataract (Eye disorders) | 1 (2) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 5 (7)
Visual disturbance (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 8 (10) | 13 (21) | 33 (37) | 6 (6) | 4 (5) | 65 (80)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 5 (6) | 5 (5) | 19 (25) | 5 (5) | 2 (4) | 37 (46)
Vomiting (Gastrointestinal disorders) | 0 (0) | 5 (5) | 4 (4) | 12 (14) | 3 (4) | 2 (6) | 26 (33)
Constipation (Gastrointestinal disorders) | 1 (2) | 2 (2) | 3 (4) | 7 (7) | 1 (1) | 3 (3) | 17 (19)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (2) | 2 (2) | 7 (7) | 2 (2) | 1 (1) | 14 (15)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 4 (4) | 0 (0) | 3 (3) | 11 (11)
Stomach discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 0 (0) | 8 (8)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Haemorrhoids (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (2) | 9 (11) | 8 (9) | 21 (24) | 2 (3) | 3 (5) | 44 (54)
Fatigue (General disorders) | 3 (3) | 6 (6) | 8 (9) | 22 (24) | 3 (5) | 0 (0) | 42 (47)
Chest pain (General disorders) | 1 (1) | 2 (2) | 3 (5) | 8 (8) | 0 (0) | 5 (6) | 19 (22)
Pyrexia (General disorders) | 0 (0) | 3 (3) | 0 (0) | 5 (5) | 3 (3) | 2 (2) | 13 (13)
Gait disturbance (General disorders) | 1 (1) | 1 (1) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 7 (8)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 6 (6)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 5 (5)
Irritability (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 10 (11) | 14 (18) | 28 (50) | 8 (11) | 12 (13) | 73 (104)
Nasopharyngitis (Infections and infestations) | 2 (3) | 3 (4) | 3 (4) | 25 (33) | 2 (2) | 3 (6) | 38 (52)
Sinusitis (Infections and infestations) | 0 (0) | 3 (7) | 6 (7) | 19 (26) | 3 (5) | 2 (2) | 33 (47)
Urinary tract infection (Infections and infestations) | 1 (3) | 5 (6) | 7 (8) | 12 (19) | 2 (3) | 3 (5) | 30 (44)
Bronchitis (Infections and infestations) | 3 (3) | 2 (2) | 7 (8) | 10 (14) | 2 (2) | 2 (2) | 26 (31)
Influenza (Infections and infestations) | 1 (1) | 5 (5) | 1 (1) | 15 (21) | 0 (0) | 2 (2) | 24 (30)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 6 (10) | 0 (0) | 3 (3) | 10 (14)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 5 (7) | 2 (2) | 0 (0) | 10 (12)
Fungal infection (Infections and infestations) | 0 (0) | 3 (4) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 6 (9)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 5 (5)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 5 (5)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 4 (6) | 14 (15) | 0 (0) | 4 (4) | 28 (31)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (4) | 8 (12) | 9 (11) | 2 (2) | 3 (3) | 24 (32)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 6 (6) | 0 (0) | 1 (1) | 9 (9)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 8 (8)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 1 (1) | 0 (0) | 7 (8)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 6 (6)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood glucose increased (Investigations) | 0 (0) | 3 (4) | 3 (4) | 10 (10) | 2 (4) | 3 (4) | 21 (26)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 2 (2) | 6 (6) | 5 (5) | 0 (0) | 1 (3) | 14 (16)
Weight increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 3 (4) | 10 (11)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 8 (10) | 1 (1) | 3 (3) | 15 (17)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 1 (1) | 4 (5) | 1 (1) | 0 (0) | 10 (11)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4) | 8 (10) | 25 (29) | 2 (2) | 3 (4) | 40 (49)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 6 (7) | 19 (26) | 1 (3) | 5 (5) | 36 (46)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (3) | 2 (3) | 7 (8) | 19 (29) | 1 (1) | 2 (2) | 32 (46)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (3) | 6 (6) | 3 (4) | 10 (12) | 1 (1) | 2 (2) | 23 (28)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 12 (13) | 0 (0) | 1 (1) | 16 (17)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 6 (7) | 1 (1) | 1 (1) | 10 (11)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 6 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 6 (6)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 6 (6)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 11 (15) | 23 (31) | 47 (59) | 9 (13) | 7 (7) | 99 (127)
Headache (Nervous system disorders) | 1 (1) | 10 (10) | 8 (15) | 31 (37) | 4 (4) | 2 (3) | 56 (70)
Tremor (Nervous system disorders) | 1 (1) | 4 (5) | 7 (8) | 21 (30) | 5 (6) | 0 (0) | 38 (50)
Balance disorder (Nervous system disorders) | 0 (0) | 2 (2) | 7 (7) | 21 (21) | 2 (3) | 5 (5) | 37 (38)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 3 (3) | 3 (4) | 15 (23) | 2 (3) | 4 (4) | 28 (38)
Somnolence (Nervous system disorders) | 0 (0) | 4 (4) | 6 (6) | 14 (15) | 0 (0) | 1 (1) | 25 (26)
Memory impairment (Nervous system disorders) | 2 (2) | 1 (1) | 4 (4) | 8 (8) | 2 (2) | 1 (1) | 18 (18)
Pallanaesthesia (Nervous system disorders) | 0 (0) | 4 (4) | 1 (2) | 8 (11) | 1 (1) | 2 (3) | 16 (21)
Amnesia (Nervous system disorders) | 2 (2) | 1 (2) | 1 (1) | 11 (13) | 1 (1) | 0 (0) | 16 (19)
Hyporeflexia (Nervous system disorders) | 0 (0) | 1 (6) | 1 (1) | 11 (17) | 1 (3) | 0 (0) | 14 (27)
Coordination abnormal (Nervous system disorders) | 0 (0) | 3 (4) | 3 (3) | 4 (4) | 0 (0) | 1 (1) | 11 (12)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 7 (7)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 5 (5)
Depression (Psychiatric disorders) | 1 (1) | 7 (7) | 3 (3) | 7 (7) | 4 (4) | 3 (3) | 25 (25)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (3) | 13 (15) | 1 (1) | 1 (1) | 19 (21)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (7) | 2 (2) | 1 (1) | 9 (12)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 5 (8) | 13 (13) | 3 (3) | 4 (5) | 27 (31)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (9) | 1 (1) | 9 (11) | 2 (3) | 0 (0) | 19 (25)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 4 (5) | 8 (9) | 1 (1) | 3 (3) | 18 (20)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4) | 2 (2) | 3 (5) | 2 (2) | 2 (2) | 11 (15)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Wound treatment (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral nerve transposition (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 4 (7) | 10 (11) | 1 (1) | 3 (4) | 21 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.